CLINICAL TRIAL: NCT03834896
Title: Madrid - Tolerance and Acceptability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY:ST2
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with dysphagia requiring Stage 1, 2 or 3 thickened fluids as determined by Speech and Language Therapist and who are expected to require provision of Stage 1, 2 or 3 thickened fluids for at least 2 further weeks.
  Interventions: Other: AYMES MADRID

INTERVENTIONS:
Other: AYMES MADRID — AYMES MADRID is a gum-based commercial thickener, that can be utilised to modify fluid consistencies to Stage 1, 2 or 3 (as per the National Descriptors for Texture Modification) to enhance the safety of fluids in those with dysphagia.

SUMMARY:
Tolerance and Acceptability of a gum based thickener.

DETAILED DESCRIPTION:
To evaluate the tolerance and acceptability of AYMES MADRID, in patients that may require modified consistency fluids. Measuring GI tolerance, compliance, convenience and preference.

To obtain data to support an ACBS submissions for AYMES MADRID (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who are able to communicate clearly.
* Patients with dysphagia requiring Stage 1, 2 or 3 thickened fluids as determined by -Speech and Language Therapist.
* Patients expected to require provision of Stage 1, 2 or 3 thickened fluids for at least 2 further weeks.
* Informed consent obtained from patient or for those without capacity following consultation with carers.

Exclusion Criteria:

* Patients with maize / corn allergy requiring a maize free diet
* Patients with inherited metabolic conditions.
* Patients requiring enteral tube feeding or parenteral nutrition.
* Patients with medical or dietary contraindication to any feed ingredients
* Patients with delayed oral phase of swallowing.
* Patients with significant renal (requiring dialysis) or hepatic impairment (e.g. hepatitis)
* Patients with dysphagia not requiring stage 1, 2 or 3 thickened fluids.
* Patients with uncontrolled inflammatory bowel disease or previous bowel resection with ongoing gastrointestinal symptoms.
* Patients for whom the investigator has concerns regarding the ability or willingness of the patient and or carer to comply with protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study (to prevent over burdening of participants and ensure a period of normalisation between study involvement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
GI side effects when using AYMES MADRID | 9 Days
  Recording of absence/presence of any nausea, vomiting, abdominal pain, bloating / flatulence, when using AYMES MADRID as assessed by presence / absence of side effect compared to baseline period.

SECONDARY OUTCOMES:
Compliance with prescription of AYMES MADRID | 9
  Recording of amount of AYMES PARIS consumed by subjects compared to amount prescribed. Good compliance = >80% of prescribed being consumed. Same data collected for baseline product and compared with that of AYMES MADRID
Bowel habits of subjects when using AYMES MADRID - frequency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES MADRID, as assessed by frequency of bowel movements (number of stools per day) and compared to same data recorded during baseline period.
Bowel habits of subjects when using AYMES MADRID - stool consistency | 9 days
  Recording of bowel habits whilst subjects consuming AYMES MADRID, as assessed by consistency of stools (assessed by Bristol Stool Chart) and compared to same data recorded during baseline period

CONTACTS AND LOCATIONS:
Locations (1):
- AYMES International Ltd., Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: No